CLINICAL TRIAL: NCT04460911
Title: Treatment Patterns And Clinical Outcomes Among Patients With Hormone Receptor-Positive/Human Epidermal Growth Factor Receptor 2-Negative Metastatic Breast Cancer (mBC) Receiving Palbociclib in Combination With Fulvestrant (PB+FUL) In The US Community Oncology Setting
Brief Title: Treatment Patterns and Clinical Outcomes Among Patients With HR+/HER2- mBC Receiving Palbociclib Combination Therapy in the US Community Oncology Setting.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481128; US oncology (Other: Alias Study Number)
Record Dates: First submitted 2020-07-06; First posted 2020-07-08 (Actual); Results first posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- PAL + FUL: Patients who initiated palbociclib-fulvestrant combination therapy as first-line or beyond therapy in the advanced or metastatic setting.

SUMMARY:
By leveraging a community-based, cancer-specific electronic healthcare record for this study, we aim to understand treatment patterns and clinical outcomes among patients with HR+/HER2- mBC who received care within the context of a large community oncology network in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of HR+/HER2- mBC
2. Initiated palbociclib + fulvestrant as first-line therapy in the metastatic setting and had at least 2 visits following the index date
3. Received care at a US oncology site(s) utilizing the full EHR at time of treatment and data are available for research purposes

Exclusion Criteria:

1. Enrollment in an interventional clinical trial during the study period
2. Evidence of prior treatment with CDK4/6 inhibitors in the metastatic setting
3. Receipt of treatment indicated for another primary cancer during the study period or history of another primary cancer documented within the US Oncology EHR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With Hormone Receptor-Positive/Human Epidermal Growth Factor Receptor 2-Negative Metastatic Breast Cancer (mBC) Receiving Palbociclib Combination Therapy, Endocrine Monotherapy Or Fulvestrant Monotherapy In The US Community Oncology Setting
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2019-10-19 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer United States, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481128

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data for participants diagnosed with hormone receptor positive (HR+)/human epidermal growth factor receptor 2 negative (HER2-) metastatic breast cancer (MBC), who initiated first line treatment with palbociclib in combination with fulvestrant between 01-February-2016 to 31-December-2019 were observed retrospectively. To allow minimum follow-up period of 6 months, participants were followed until 30 June 2020, last participant record or date of death, whichever occurred first.
Pre-assignment Details: Data was retrieved from electronic healthcare record (EHR) and available data was evaluated over 2.5 years of this retrospective observational study.
Groups:
- Palbociclib + Fulvestrant: Participants who initiated palbociclib in combination with fulvestrant as first line therapy for HR+/HER2- MBC during the period 01-February-2016 to 31-December-2019 were included in this retrospective observational study. Participants were followed up until 30-Jun-2020.
Period: Overall Study
Arm/Group | Palbociclib + Fulvestrant
Started | 317
Completed | 317
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Arm/Group | Palbociclib + Fulvestrant
Number analyzed (Participants) | 317
Age, Continuous [Median (Full Range); unit: Years] | 67.3 [34.5 to 93.5]
Age, Customized [Count of Participants; unit: Participants]
  18-50 | 22
  51-70 | 174
  More than (>) 70 | 121
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 312
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 27
  Not documented | 41
  Other | 10
  White | 239
Body Mass Index (BMI) at Index Date [Mean (Standard Deviation); unit: Kilogram per square meter] | 28.8 (6.9)
Number of Participants According to Smoking history [Count of Participants; unit: Participants] — Number of participants classified according to smoking history were reported.
  Participants
    Never smoked | 111
    Current smoker | 18
    Former smoker | 81
    No information | 107
Number of Participants According to Family History of Cancer [Count of Participants; unit: Participants] — Number of participants classified according to family history of cancer were reported.
  Participants
    Yes | 206
    No/no information | 111
Number of Participants According to Menopausal Status [Count of Participants; unit: Participants] — Number of participants classified according to menopausal status were reported.
  Participants
    Pre-menopausal | 9
    Peri-menopausal | 1
    Post-menopausal | 287
    No information | 20
Time Since Initial BC Diagnosis [Mean (Standard Deviation); unit: Weeks] — The duration of time, in weeks, between the date of BC diagnosis and presentation of metastatic disease were reported. Population: Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
  Weeks
    number analyzed (Participants) | 316
    (all) | 380.6 (328.3)
Time Since MBC Diagnosis [Mean (Standard Deviation); unit: Weeks] — The duration of time, in weeks, between the index date and presentation of metastatic disease were reported. Index date was defined as the date of the first administration of either drug (palbociclib or fulvestrant).
  Weeks | 7.5 (34.0)
Number of Participants According to Distant Metastatic Sites [Count of Participants; unit: Participants] — Number of participants classified according to the distant metastatic sites were reported. No information signifies that metastases were not documented in the chart, not necessarily that participants did not have metastases. One participant may have more than 1 sites of metastasis.
  Participants
    Bone (single) | 47
    Bone (multiple) | 181
    Brain | 8
    Liver (single) | 19
    Liver (multiple) | 43
    Lung (single) | 28
    Lung (multiple) | 41
    Lung (pleural effusion) | 36
    Lymph nodes (regional) | 32
    Lymph nodes (distant) | 43
    Ovary | 1
    Other | 47
Number of Participants According to Disease-Free Interval [Count of Participants; unit: Participants] — Disease-free interval was defined as the duration between discontinuation of adjuvant therapy and the start of treatment for metastatic disease. Population: Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
  Participants
    Less than (<) 12 months: number analyzed (Participants) | 269
    Less than (<) 12 months | 178
    More than or equal to (>=) 12 months: number analyzed (Participants) | 269
    More than or equal to (>=) 12 months | 91
Number of Participants According to Visceral/non-Visceral Status [Count of Participants; unit: Participants] — Number of participants classified according to visceral or non-visceral status were reported.
  Participants
    Asymptomatic visceral disease | 105
    Bone only | 117
    Non-visceral disease | 27
    Not documented | 14
    Other | 5
    Symptomatic visceral disease | 49
Number of Participants According to Count of Metastatic Sites [Count of Participants; unit: Participants] — Number of participants classified according to the count of metastatic sites were reported.
  Participants
    1 | 178
    2 | 83
    3 | 44
    4+ | 12
Number of Participants According to Stage at Diagnosis [Count of Participants; unit: Participants] — Tumor Node Metastasis(TNM): based on tumor size, metastasis to nearby lymph nodes(LN),or distant metastasis. Stages were: stage 0(no evidence of cancer cells),stage 1(T1N0M0),stage IA(T1N0M0),stage IB(T0 or T1N1M0),stage IIA(T0N1M0,T1N1M0,T2N0M0),stage IIB(T2N1M0,T3N0M0),stage IIIA(T0N2M0,T1N2M0,T2N3M0,T3N1 or N2M0),stage IIIB(T4 any NM0,any TN3M0),stage IIIC(any TN3M0),stage IV(any T any NM1),where T0=early form of tumor,T1= <2 centimeter(cm),T2=2-5 cm,T3= >2 cm,T4=large sized,N0=not spread to LN,N1=spread to 1 to 3,N2=spread to 4 to 9,N3=spread >10 axillary LN,M0=no metastasis,M1=metastasis.
  Participants
    Stage I | 0
    Stage IA | 18
    Stage IB | 3
    Stage IIA | 33
    Stage IIB | 31
    Stage IIIA | 26
    Stage IIIB | 4
    Stage IIIC | 12
    Stage IV | 41
    No information | 149
Number of Participants According to Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG performance status score is a rating of a participant's disease status, daily living activities and quality of life, where 0 indicates fully active,1 indicates restricted in physically strenuous activity, 2 indicates ambulatory and capable of self-care but unable to work, 3 indicates capable only of limited self-care, 4 indicates completely disabled and 5 indicates dead. Higher scores indicated more severe disease, difficulty in performing daily activity and poor quality of life. Number of participants classified according to ECOG performance status.
  Participants
    0 | 73
    1 | 107
    2 | 26
    More than or equal to (>=) 3 | 5
    Not documented | 106
Number of Participants According to Comorbidities [Count of Participants; unit: Participants] — Number of participants classified according to comorbidities documented within 6 months prior to or on index date were reported. Index date was defined as the date of the first administration of either drug (palbociclib or fulvestrant). Population: Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
  Participants
    Atrial fibrillation: number analyzed (Participants) | 306
    Atrial fibrillation | 6
    Cerebrovascular disease: number analyzed (Participants) | 306
    Cerebrovascular disease | 3
    Congestive heart failure: number analyzed (Participants) | 306
    Congestive heart failure | 4
    Chronic pulmonary disease: number analyzed (Participants) | 306
    Chronic pulmonary disease | 15
    Connective tissue disease: number analyzed (Participants) | 306
    Connective tissue disease | 3
    Dementia: number analyzed (Participants) | 306
    Dementia | 2
    Diabetes with end organ damage: number analyzed (Participants) | 306
    Diabetes with end organ damage | 10
    Diabetes without end organ damage: number analyzed (Participants) | 306
    Diabetes without end organ damage | 38
    Depression: number analyzed (Participants) | 306
    Depression | 29
    Human Immunodeficiency Virus/Acquired Immunodeficiency Syndrome(HIV/AIDS): number analyzed (Participants) | 306
    Human Immunodeficiency Virus/Acquired Immunodeficiency Syndrome(HIV/AIDS) | 1
    Hypertension: number analyzed (Participants) | 306
    Hypertension | 112
    Infection: number analyzed (Participants) | 306
    Infection | 1
    Long QT syndrome (drug induced): number analyzed (Participants) | 306
    Long QT syndrome (drug induced) | 1
    Mild liver disease: number analyzed (Participants) | 306
    Mild liver disease | 2
    Moderate to severe renal disease: number analyzed (Participants) | 306
    Moderate to severe renal disease | 9
    Myocardial infarction: number analyzed (Participants) | 306
    Myocardial infarction | 3
    Peptic ulcer disease: number analyzed (Participants) | 306
    Peptic ulcer disease | 2
    Peripheral vascular disease: number analyzed (Participants) | 306
    Peripheral vascular disease | 1
    Tachycardia: number analyzed (Participants) | 306
    Tachycardia | 1
    Stroke: number analyzed (Participants) | 306
    Stroke | 3
    Venous thromboembolism (pulmonary embolism or deep vein thrombosis): number analyzed (Participants) | 306
    Venous thromboembolism (pulmonary embolism or deep vein thrombosis) | 13
    Hypotension: number analyzed (Participants) | 306
    Hypotension | 47
Number of Participants According to Disease Histology [Count of Participants; unit: Participants] — Number of participants classified according to disease histology were reported.
  Participants
    Ductal | 142
    Lobular | 27
    Other | 3
    No information | 145
Number of Participants According to Breast Cancer Gene (BRCA) 1/2 Status [Count of Participants; unit: Participants] — Number of participants classified according to Breast cancer gene (BRCA) 1/2 status were reported.
  Participants
    Positive | 4
    Negative | 27
    Not documented | 286
Number of Participants According to Estrogen Receptor 1 Gene (ESR1) Status [Count of Participants; unit: Participants] — Number of participants classified according to Estrogen receptor 1 gene (ESR1) status were reported.
  Participants
    Positive | 1
    Negative | 7
    Not documented | 309
Number of Participants According to Next Generation Sequencing (NGS) Status [Count of Participants; unit: Participants] — Number of participants classified according to Next generation sequencing (NGS) status were reported.
  Participants
    Positive | 7
    Negative | 5
    No information | 305

OUTCOME MEASURES:

1. Primary Outcome: Time to Chemotherapy
Description: Time to chemotherapy was defined as the interval (in weeks) between index treatment (palbociclib +fulvestrant) and start of chemotherapy as documented in the iKnowMed (iKM) EHR database. Participants with ongoing treatment at the study observation period were censored on the study end date or the last visit date available in the dataset, whichever occurred first. Kaplan-Meier method was used for analysis.
Time Frame: From start of index treatment until start of chemotherapy or censoring date, during study observation period maximum up to approximately 53 months (data was retrieved and observed during 2.5 years of this retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Palbociclib + Fulvestrant
Number analyzed (Participants) | 317
Weeks | NA [33.5 to NA] — Median and upper limit of 95% CI was not estimable due to Iess number of participants with an event.

2. Primary Outcome: Number of Participants According to Reasons for Treatment Discontinuation
Description: The number of participants classified according to the reasons for treatment discontinuation were reported in this outcome measure.
Time Frame: From start of index treatment until stop of index treatment or censoring date, during study observation period maximum up to approximately 53 months (data was retrieved and observed during 2.5 years of this retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Fulvestrant
Number analyzed (Participants) | 250
Participants
  Provider-documented disease progression | 133
  Death | 20
  Insurance/cost-related | 1
  Patient preference | 15
  Toxicity | 44
  Other | 17
  No information | 20

3. Primary Outcome: Real-World Duration of Treatment (rwDOT)
Description: Real-world duration of treatment (rwDOT) was defined as the interval between the start and stop index treatment as documented in the iKM EHR database. Participants with ongoing treatment at the study observation period were censored on the study end date or the last visit date available in the dataset, whichever occurred first. Kaplan-Meier method was used for analysis.
Time Frame: as for outcome 2
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Palbociclib + Fulvestrant
Number analyzed (Participants) | 317
Weeks | 15.8 [13.7 to 18.4]

4. Primary Outcome: Time to Next Treatment (TTNT) From Index Treatment
Description: Time to next treatment (TTNT) was defined as the interval between the start of the index treatment and the date of the next-line treatment as documented in the iKM EHR database. Participants who did not advance to the next treatment within the study observation period were censored on the study end date or the last visit date available in the dataset, whichever occurred first. Kaplan-Meier method was used for analysis.
Time Frame: From start of index treatment to date of next line treatment or censoring date, during study observation period maximum up to approximately 53 months (data was retrieved and observed during 2.5 years of this retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Palbociclib + Fulvestrant
Number analyzed (Participants) | 317
Weeks | 16.8 [14.7 to 22.0]

5. Primary Outcome: Percentage of Participants With Provider Documented Disease Progression
Description: Percentage of participants with provider documented progression (documented as disease has progressed or worsening of disease) is reported in this outcome measure.
Time Frame: From start of treatment until documented disease progression, during study observation period maximum up to approximately 53 months (data was retrieved and observed during 2.5 years of this retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Fulvestrant
Number analyzed (Participants) | 317
Percentage of participants | 42.0

6. Primary Outcome: Real-World Time to Tumor Progression (rwTTP)
Description: The rwTTP was measured from the initiation of index treatment to the date of provider-documented progression (documented by provider as disease has progressed or worsening of disease), censoring participants without evidence of provider-documented progression at the last visit date. Kaplan-Meier method was used for analysis.
Time Frame: From initiation of the index treatment to the date of progression or censoring date, during study observation period maximum up to approximately 53 months (data was retrieved and observed during 2.5 years of this retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Palbociclib + Fulvestrant
Number analyzed (Participants) | 317
Weeks | 26.7 [21.6 to 34.7]

7. Primary Outcome: Real-World Progression-Free Survival (rwPFS)
Description: The rwPFS was measured from the initiation of the index treatment to the date of progression (documented by provider as disease has progressed or worsening of disease) or date of death due to any cause, censoring participants who were still alive at the end of the study observation period and did not progress at the last visit date. Kaplan-Meier method was used for analysis.
Time Frame: From initiation of index treatment to date of progression or death due to any cause or censoring date, during study observation period maximum up to approximately 53 months (data was retrieved and observed during 2.5 years of this retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Palbociclib + Fulvestrant
Number analyzed (Participants) | 317
Weeks | 19.6 [15.2 to 23.6]

8. Primary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the interval between index treatment and the date of death (any cause) as documented in the Limited Access Death Master File (LADMF), National Death Index (NDI) and the iKM EHR database. Participants who did not die within the study observation period were censored on the study end date or the last visit date available in the dataset, whichever occurred first. Kaplan-Meier method was used for analysis.
Time Frame: From start of index treatment until date of death or censoring date, during study observation period maximum up to approximately 53 months (data was retrieved and observed during 2.5 years of this retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Palbociclib + Fulvestrant
Number analyzed (Participants) | 317
Weeks | 44.1 [39.4 to NA] — Upper limit of 95% CI was not estimable due to Iess number of participants with an event.

9. Other Pre Specified Outcome: Percentage of Participants According to the Dosing Strength of Fulvestrant and Palbociclib as Their Index Treatment
Description: The percentage of participants classified according to the dosing strength of Palbociclib and Fulvestrant as their index treatment were reported in this outcome measure. Index date was the date of initiation with palbociclib + fulvestrant during the study identification period.
Time Frame: At index, anytime between 01-February-2016 and 31-December-2019 (data was retrieved and observed during 2.5 years of this retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Fulvestrant
Number analyzed (Participants) | 317
Percentage of participants
  Fulvestrant at 500 Milligram (mg) | 93.4
  Palbociclib at 125 mg | 92.4

10. Other Pre Specified Outcome: Duration of Treatment for Advanced Metastatic Breast Cancer
Description: The duration of treatment for advanced metastatic breast cancer was reported in this outcome measure.
Time Frame: From start of index treatment until stop of index treatment, during study observation period maximum up to approximately 53 months (data was retrieved and observed during 2.5 years of this retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Palbociclib + Fulvestrant
Number analyzed (Participants) | 317
Weeks | 44.7 [0 to 227.6]

11. Other Pre Specified Outcome: Percentage of Participants With Prior Adjuvant Hormonal Treatment for Advanced Metastatic Breast Cancer
Description: Percentage of participants with prior adjuvant hormonal treatment for breast cancer were reported in this outcome measure. Index date was the date of initiation with palbociclib + fulvestrant during the study identification period.
Time Frame: Prior to index date (the date of initiation with Palbociclib-Fulvestrant during the study identification period) (data was retrieved and observed during 2.5 years of this retrospective study)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Fulvestrant
Number analyzed (Participants) | 254
Percentage of participants | 43.7

12. Other Pre Specified Outcome: Number of Participants According to Year of Treatment Initiation for Advanced Metastatic Breast Cancer
Description: Number of participants were classified according to the year of treatment initiation for advanced metastatic breast cancer in this outcome measure.
Time Frame: Quarter(Q)1 2015,Q2 2015,Q3 2015,Q4 2015,Q1 2016,Q2 2016,Q3 2016,Q4 2016,Q1 2017,Q2 2017,Q3 2017,Q4 2017,Q1 2018,Q2 2018,Q3 2018,Q4 2018,Q1 2019,Q2 2019,Q3 2019,Q4 2019(data was retrieved and observed during 2.5 years of this retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Fulvestrant
Number analyzed (Participants) | 317
Participants
  Quarter (Q) 1 2015 | 0
  Q2 2015 | 0
  Q3 2015 | 0
  Q4 2015 | 0
  Q1 2016 | 10
  Q2 2016 | 12
  Q3 2016 | 8
  Q4 2016 | 18
  Q1 2017 | 17
  Q2 2017 | 24
  Q3 2017 | 30
  Q4 2017 | 31
  Q1 2018 | 23
  Q2 2018 | 21
  Q3 2018 | 15
  Q4 2018 | 18
  Q1 2019 | 18
  Q2 2019 | 25
  Q3 2019 | 20
  Q4 2019 | 27

13. Other Pre Specified Outcome: Percentage of Participants With Change in Dose
Description: The percentage of participants with dose change for index treatment were reported in this outcome measure.
Time Frame: From index treatment until follow up period of 6 months (data was retrieved and observed during 2.5 years of this retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib + Fulvestrant
Number analyzed (Participants) | 317
Percentage of participants
  Yes | 77.6
  No change/no documentation | 22.4

ADVERSE EVENTS:
Time Frame: For adverse events, not applicable as adverse events were not collected during the study. For all-cause mortality, from start of index treatment until end of study observation period maximum up to approximately 53 months (data was retrieved and observed during 2.5 years of this retrospective study).
Description: This observational retrospective study retrieved data from medical records and the data existed as unstructured data. In these data sources, individual participant data were not retrieved or validated, and it was not possible to link a particular product and medical event for any individual. Thus, the minimum criteria (identifiable participant, identifiable reporter, a suspect product, and event) for reporting an adverse event could not be met, hence safety data were not collected and reported.
Arm/Group | Palbociclib + Fulvestrant
All-Cause Mortality (participants affected / at risk) | 92/317
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/11/NCT04460911/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT04460911/SAP_001.pdf